CLINICAL TRIAL: NCT01798303
Title: Multicenter, Randomized, Double-Blind, Parallel-Group, Placebo-Controlled Trial in Patients With Alcohol Dependence
Brief Title: A Study of LY2940094 in Participants With Alcohol Dependency
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BlackThorn Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14792; I5J-MC-NOAD (Other: Eli Lilly and Company)
Record Dates: First submitted 2013-02-21; First posted 2013-02-25 (Estimated); Last update posted 2017-02-03 (Estimated); Status verified 2017-02

CONDITIONS: Alcoholism
MeSH Terms: conditions — Alcoholism | interventions — LY2940094

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- LY2940094 (Experimental): 40 mg LY2940094 oral tablet, QD for 8 weeks
  Interventions: Drug: LY2940094
- Placebo (Placebo Comparator): Identically matched placebo oral tablet, QD for 8 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY2940094 — Administered orally
  Arms: LY2940094
Drug: Placebo — Administered orally
  Arms: Placebo

SUMMARY:
The main purpose of this study is to evaluate a once daily (QD) 40-milligram (mg) oral dose of LY2940094 in participants with an alcohol dependency to evaluate if LY2940094 will reduce alcohol drinking in these participants. The study will last for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Present with alcohol dependence (AD) defined by the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision (DSM-IV-TR 303.9)
* Must have 3 to 6 heavy drinking days per week as assessed by the Timeline Follow Back (TLFB) scale at screening and baseline (heavy drinking is defined as greater than 4 drinks per day for females and greater than 5 drinks per day for males)
* Have a body mass index (BMI) between 18 and 35 kilograms per square meter (kg/m^2)

Exclusion Criteria:

* Have had prior seizures or other condition that would place the participant at increased risk of seizures, and participants taking anticonvulsants for seizure control
* Have any other clinically significant medical condition or circumstance prior to randomization that, in the opinion of the investigator, could affect participant safety
* Meet Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, (DSM-IV) Axis I criteria for a lifetime diagnosis of schizophrenia, schizoaffective disorder, bipolar I disorder, or other psychoses

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2013-07; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Change from Baseline to Week 8 in the Average Number of Drinks per Day (NDD) Measured Over 28 Days | Baseline, Week 8

SECONDARY OUTCOMES:
Change from Baseline to Week 8 in Gammaglutamyl Transferase (GGT) | Baseline, Week 8
Percentage of Heavy Drinking Days per Month | Baseline and Week 8
Percentage of Days Abstinent per Month | Baseline and Week 8
Percentage of Participants with No (0) Heavy Drinking Days per Month | Baseline and Week 8

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST, Study Director — Eli Lilly and Company
Locations (5):
- United States (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New Haven, Connecticut
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., North Miami, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Indianapolis, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Portland, Oregon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Charleston, South Carolina